CLINICAL TRIAL: NCT04909892
Title: A Phase 2a Study of Intravenous Allogeneic Adipose-Derived Mesenchymal Stem Cells to Treat Post COVID-19 "Long Haul" Pulmonary Compromise
Brief Title: Study of Allogeneic Adipose-Derived Mesenchymal Stem Cells to Treat Post COVID-19 "Long Haul" Pulmonary Compromise
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Replaced by a different protocol.
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC-PLH-201
Record Dates: First submitted 2021-05-29; First posted 2021-06-02 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: covid-19; long haul; post-acute covid
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COVI-MSC 1 vial (Experimental): Subjects will receive intravenous infusions of COVI-MSC (one vial, ~18.5 million cells) on Day 0, Day 2, and Day 4.
  Interventions: Biological: COVI-MSC
- COVI-MSC 2 vials (Experimental): Subjects will receive intravenous infusions of COVI-MSC (two vials, ~37 million cells) on Day 0, Day 2, and Day 4.
  Interventions: Biological: COVI-MSC

INTERVENTIONS:
Biological: COVI-MSC — COVI-MSC are allogeneic culture-expanded adipose-derived mesenchymal stem cells

SUMMARY:
This is a Phase 1b study to assess the safety and efficacy of COVI-MSC in treating post COVID-19 "long haulers" with pulmonary compromise.

DETAILED DESCRIPTION:
This is a Phase 1b multicenter study to assess the safety and efficacy of COVI-MSC in treating post COVID-19 "long haulers" with pulmonary compromise.

COVI-MSC will be administered intravenously on Day 0, Day 2, and Day 4.

ELIGIBILITY:
Inclusion Criteria:

* Has had prior laboratory-confirmed SARS-CoV-2 infection as determined by an approved polymerase chain reaction (PCR) or an approved antigen test of any specimen
* Has had a recent (within a week) negative SARS-CoV-2 test (an approved PCR or antigen test)
* Has had at least moderate or severe post-COVID-19 pulmonary symptoms for at least 3 months which have resulted in reduced physical functioning compared to pre-COVID-19 status
* Willing to follow contraception guidelines

Exclusion Criteria:

* Clinically improving pulmonary status over the month prior to screening
* Undergone a previous stem cell infusion unrelated to this trial
* Pregnant or breast feeding or planning for either during the study
* Suspected uncontrolled active bacterial, fungal, viral, or other infection
* History of a splenectomy, lung transplant or lung lobectomy
* Concurrent participation in another clinical trial involving therapeutic interventions (observational study participation is acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change in 6-Minute Walk Distance (6MWD) at Day 60 | Baseline to Day 60
  Change in 6MWD at Day 60

SECONDARY OUTCOMES:
Change in 6MWD at Day 30 | Baseline to Day 30
  Change in 6MWD at Day 30
Change in Pulmonary Function Tests (PFTs) | Baseline to Day 30 and Day 60
  Change in PFTs at Days 30 and 60, as assessed using Forced Vital Capacity, Forced Expiratory Volume, Total Lung Capacity, and diffusing capacity for carbon monoxide (DLCO)
Change in oxygenation | Baseline to Day 30 and Day 60
  Change in oxygenation at Days 30 and 60, as measured using SpO2/FiO2 ratio
Change in biomarker levels | Baseline through Day 30
  Change in biomarker levels: plasma lipocalcin-2, matrix metalloproteinase-7, hepatocyte growth factor

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.